CLINICAL TRIAL: NCT06962592
Title: A Community-based Adaptation of a Peer-led Intervention to Address Alcohol Use and HIV Risk in Pregnant Women in South Africa (Mentor Moms+)
Brief Title: Mentor Moms+ Study
Acronym: (MM+)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of Cape Town (Other); San Diego State University (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Dvora Joseph Davey, PhD, MPH, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 24-0130; R34AA030942 (NIH)
Record Dates: First submitted 2025-04-08; First posted 2025-05-08 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: HIV; Alcohol Consumption
Keywords: pregnant; postpartum; HIV prevention; HIV treatment; Alcohol use; breastfeeding
MeSH Terms: conditions — Alcohol Drinking; Breast Feeding

STUDY DESIGN:
Intervention Model Description: For the pilot RCT, we will randomize enrolled, consented participants into one of two study arms, MM+ intervention or enhanced HIV attention control, in a 1:1 ratio.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MM+ Intervention (Experimental): MM+ will involve mentor mother delivery of brief MI sessions individually over a series of clinic- based visits over a 6m period during pregnancy and postpartum. Intervention content, duration, and full menu of HIV prevention services offered will be finalized prior to launch. We anticipate no fewer than five to six 15-20 minute MI sessions focused on the benefits of reducing alcohol use during pregnancy, managing HIV risk among women without HIV and importance of ART use and viral suppression for reducing the risk of vertical transmission. Participants in MM+ arm will receive enhanced HIV prevention counseling integrated into routine antenatal care visits, including PrEP and ART biofeedback adherence counseling, provided by a trained study nurse. Participants in the intervention arm will also receive EtG testing (alcohol use) and corresponding biofeedback counseling.
  Interventions: Behavioral: MM+
- Enhanced HIV attention control (eSOC) (Active Comparator): Similar to placebo pills, attention control is often used in randomized trials for behavioral interventions to control for the nonspecific effects of the intervention. Given that existing MM models focus on prevention of vertical transmission and HIV treatment and our primary interest is understanding how inclusion of alcohol reduces alcohol use improves adoption of ART/PrEP use, we will use an enhanced HIV attention control with the same time frame for the intervention (e.g. 2-3 sessions during antenatal/and 2-3 sessions during postpartum periods). Sessions will consist of educational counseling on HIV risk, partner testing modalities as well as PrEP/ART urine assay testing followed by real-time in-clinic adherence counseling delivered privately by lay counselors (different from MM+ arm to avoid contamination), all coinciding with routine ANC visits when possible.
  Interventions: Behavioral: Enhanced HIV attention control (eSOC)

INTERVENTIONS:
Behavioral: MM+ — Participants in both study arms will receive clinic-based HIV counseling, including urine tenofovir testing and biofeedback counseling on recent PrEP or ART use. Activities unique to women enrolled in the intervention arm include: Brief motivational interviewing sessions with a mentor mother focusing on 1) EtG testing and biofeedback on recent alcohol use, 2) counseling and mentorship on ways to reduce alcohol use.
  Arms: MM+ Intervention
Behavioral: Enhanced HIV attention control (eSOC) — Participants in the enhanced HIV attention control arm (comparison group) will attend a similar number of study visits within the same time frame as intervention participants (5-6 sessions during 6-month timeframe including both pregnancy and postpartum). Control arm sessions will consist of one-on-one educational counseling on HIV risk, partner HIV testing modalities, as well as conducting PrEP/ART urine assay testing followed by real-time in-clinic adherence counseling delivered privately (different from study nurses delivering PrEP/ART biofeedback in MM+ intervention arm to avoid contamination), all coinciding with routine ANC visits.
  Arms: Enhanced HIV attention control (eSOC)

SUMMARY:
The goal of this study is to adapt an existing evidence based intervention for use in pregnant and lactating people (PLP) who use alcohol. Through the pilot RCT, we aim to understand if tailored intervention, Mentor Mothers+, is effective in reducing alcohol use (primary outcome) and improving antiretroviral (PrEP or ART) adherence (secondary outcomes) among pregnant and breastfeeding women living with and without HIV in a community heavily burdened by this syndemic.

The investigators will conduct an pilot randomized control trial in 100 pregnant women, recruited during antenatal care (ANC) visits within the Saldanha Bay Municipality clinic in Cape Town, South Africa. The RCT will involve the delivery of brief, individual motivational interviewing sessions provided by trained mentor mothers from the community who are on either PrEP (living without HIV) or ART (living with HIV) and who stopped or reduced alcohol use during pregnancy. The enrolled participants will be followed for a 6-month period spanning both pregnancy and postpartum stages.

DETAILED DESCRIPTION:
The syndemic of alcohol use and HIV risk in pregnant and lactating people (PLP) threatens the health of mother, fetus, children and families in South Africa. PLP living with HIV who use alcohol may access antiretroviral therapy (ART) late or disengage with ART care, increasing the risk of vertical HIV transmission. PLP not living with HIV who use alcohol are at increased risk of HIV and may require targeted interventions to receive pre-exposure prophylaxis (PrEP) delivery and adherence counselling. Alcohol use also increases risk of HIV acquisition and poor ART adherence. The "mentor mother" (MM) intervention model is an evidence-based intervention (EBI) with demonstrated success in improving HIV and antenatal care outcomes. The model utilizes a task-shifting approach; positive deviant peers (mothers) deliver interventions to PLP within and outside of the antenatal clinic.

Our study aims to evaluate the feasibility and acceptability of MM+ on reduction of alcohol use (primary outcome) and PrEP use (in PLP without HIV) and ART adherence (in PLP living with HIV) (secondary outcomes) in a pilot randomized control trial (RCT) in n=100 pregnant women who currently use alcohol. Primary outcome: Reduced alcohol use following the intervention (at 6m via phosphatidylethanol [PEth] levels). Secondary outcomes: PrEP and ART continued use at 6 months via urine tenofovir levels at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* • ≥ 16 years;

  * Pregnancy confirmed;
  * reported alcohol use during pregnancy (in last 2 months);
  * lives within 20 kilometers of the study facility;
  * able and willing to consent to study participation.

Exclusion Criteria:

* Individuals not meeting the above criteria will be excluded.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Reduction in alcohol use (objective) | From enrollment to the end of intervention period at 6 months
  Reduced alcohol use following the intervention delivery, measured via:dried blood spot (DBS) testing of phosphatidylethanol (PEth) levels
  Alcohol consumption via PEth will be defined as <20 ng/mL representing light or no consumption, >20-<200 ng/mL indicating consumption and ≥200ng/mL indicating significant or heavy recent alcohol use in past 21 days.
Reduction in alcohol use (self-report) | From enrollment to the end of intervention period at 6 months
  Reduced alcohol use following the intervention delivery,measured via: self-report (AUDIT-C score).
  Self-reported alcohol use (via participant survey) will be categorically defined via AUDIT-C score of 0 indicating abstinence versus score >0 indicating recent alcohol use.

SECONDARY OUTCOMES:
PrEP Initiation | From enrollment to the end of intervention period at 6 months
  Initiation to PrEP evaluated via patient medical records
PrEP Adherence | From enrollment to the end of intervention period at 6 months
  Adherence to PrEP evaluated via urine tenofovir testing results
ART Adherence | From enrollment to the end of intervention period at 6 months
  Adherence to ART measured via urine tenofovir (TFV) testing results. Urine TFV results will reflect recent ART adherence (past 48-72 hours).
ART Adherence | From enrollment to the end of intervention period at 6 months
  Adherence to ART measured via participant self-report
HIV Viral Load | From enrollment to the end of intervention period at 6 months
  HIV viral load levels will be evaluated among participants living with HIV and on ART

CONTACTS AND LOCATIONS:
Locations (2):
- South Africa (2):
  - Saldanha Bay Municipality Clinic, Cape Town, Western Cape
  - Saldanha Bay Clinics, Saldanha Bay, Western Cape

IPD SHARING:
Plan to Share IPD: Yes
The study team will share de-identified data upon request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1 year following study start through 1 year following study end
Access Criteria: Email PI with full request: dvoradavey@ucla.edu

REFERENCES:
- [Derived] Essack Z, Petersen Z, Miller AP, Schoetz Dean S, Daniels D, Hofmeester H, Belin T, van Rooyen H, Louw J, Joseph Davey D. Community-Based Adaptation and Evaluation of a Peer-Led Intervention to Address Alcohol Use and HIV in Pregnant and Breastfeeding Women in South Africa: Protocol for the "Mentor Mothers Plus" Randomized Control Trial. JMIR Res Protoc. 2025 Dec 18;14:e78856. doi: 10.2196/78856. PMID 41411648